CLINICAL TRIAL: NCT01606475
Title: Human Alloislet Transplant for Type 1 or Surgical Diabetes Mellitus With Complications
Brief Title: Islet Transplant for Type 1 or Surgical Diabetes
Acronym: EXAX
Status: No longer available | Type: Expanded Access
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1108M03061
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia; Labile Diabetes; End-stage Renal Disease
Keywords: Islet transplant; Diabetes Mellitus; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Kidney Failure, Chronic; Diabetes Mellitus

INTERVENTIONS:
Biological: Allogeneic islets of Langerhans — Up to 3 intraportal infusions of cadaveric pancreatic islets of Langerhans. Each infusion to contain at least 5,000 islet equivalents/kg body weight.
  Other Names: Islets

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of islet transplants from human cadaver donors into type 1 or surgical diabetes mellitus patients who experience frequent acute or advanced chronic complications but do not qualify for other islet transplant trials. Under this protocol, patients may receive intraportal alloislet transplant under one of the following scenarios:

1. islet transplant alone
2. simultaneous islet-kidney transplant, or 3)islet after kidney transplant.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the efficacy of islet allotransplants for labile diabetes mellitus in patients who do not meet standard inclusion/exclusion criteria for any other islet transplant trials in the US and are not good candidates for a pancreas transplant. We expect that this will include patients who have surgical diabetes (total pancreatectomy) rather than type 1 diabetes, patients who are highly sensitized (PRA>20%), and patients who have had prior failed pancreas transplantation. These patients may have equally severe hypoglycemia, glucose lability, and/or severe microvascular complications, but are excluded from standard islet transplant trials currently available in the U.S.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 18 to 70 years of age.
2. Ability to provide written informed consent.
3. Mentally stable and able to comply with the procedures of the study protocol.
4. Insulin-dependent diabetes mellitus
5. Not otherwise eligible for an existing alloislet transplant protocol for type 1 diabetes mellitus
6. Involvement in intensive diabetes management, defined by at least 3 injections daily or insulin pump therapy.
7. Meets at least one of the following criteria despite intensive efforts made in close cooperation with their diabetic care team:

   * Significant hypoglycemia unawareness or glycemic lability on conventional insulin therapy, as evidenced by at least one of the following at screening:
   * Clarke score > 4
   * HYPO score >90th percentile (1047)
   * Lability index (LI) >90th percentile (433 mM2/h/wk)
   * A composite of a Clarke score of 4 or more and a HYPO score greater than or equal to the 75th percentile (423) and a LI greater than of equal to the 75th percentile (329)
   * Progressive secondary complications as defined by end-stage renal disease necessitating dialysis or renal transplantation (eligible for islet after kidney or simultaneous islet kidney transplant) AND islet transplant appears to provide a more satisfactory benefit to risk ratio compared to pancreas transplantation (eg high surgical risk)

Exclusion Criteria:

1. HbA1c >10%.
2. Untreated proliferative diabetic retinopathy.
3. Uncontrolled Hypertension (SBP>160 or DBP>100)
4. For female participants: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study.
5. Active infection including hepatitis B, hepatitis C, HIV, or TB as determined by a positive skin test or clinical presentation, or under treatment for suspected TB.
6. Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin.
7. Receiving treatment for a medical condition requiring chronic use of systemic steroids, except for use of prednisone <5 mg per day for kidney transplant recipients or physiologic hydrocortisone replacement.
8. Persistent elevation of liver function tests at the time of study entry. Persistent SGOT (AST), SGPT (ALT), Alk Phos or total bilirubin, with values >1.5 times normal upper limits will exclude a patient.
9. Severe co-existing cardiac disease, characterized by any one of these conditions:

   * recent myocardial infarction (within past 6 months).
   * evidence of ischemia on functional cardiac exam within the last year.
   * left ventricular ejection fraction <30%.
10. If diabetes is secondary to total pancreatectomy, participants will be considered only if >1 year out from surgery, medically stable, without severe issues with bowel function or pain management that may interfere with safe completion of the trial.
11. History of alcoholism
12. Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard J Hering, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States